

## **Consent Form**

Feasibility and Acceptability of Body Signal Integration Training for functional neurological disorder: A case series



## **Consent Form**

## Feasibility and Acceptability of Body Signal Integration Training for functional neurological disorder: A case series

If you are happy to participate, please complete and sign the consent form below.

| | Activities | Initials |
|---|---|---|
| 1 | I confirm that I have read the attached information sheet (Version 5: 08.02.23) for the above study and have had the opportunity to consider the information and ask questions and had these answered satisfactorily. | |
| 2 | I understand that my participation in the study is voluntary and that I am free to withdraw at any time without giving a reason and without detriment to myself. I understand that if I drop out at any point, researchers will retain any information gathered unless I specifically request that it be destroyed. | |
| | I agree to take part on this basis. | |
| 3 | I agree to therapy sessions being video recorded for the purpose of Clinical Supervision | |
| 4. | I consent to provide contact details for my GP so that a standardised letter can be sent to my GP to inform them of my participation in the study. | |
| 5. | I agree that any data collected may be included in anonymous form in publications and conference presentations. | |
| 6. | I understand that data collected during the study may be looked at by individuals from The University of Manchester or regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my data. | |
| 7. | I understand that my full name and email address will be passed to the University's Finance team for the sole purpose of sending me the shopping voucher. | |
| 8. | I understand that there may be instances where during the course of the research information is revealed which means the researchers will be obliged to break confidentiality and this has been explained in more detail in the information sheet. | |
| 9. | I agree to take part in this study. | |

The following activities are optional, you may participate in the research without agreeing to the following:



| 10. | I agree that any anonymised data from questionnaires collected may be made available to other researchers |
|---|---|
| 11. | I agree that the researchers may contact me in future about other research projects. |
| 12. | I agree that the researchers may retain my contact details in order to provide me with a summary of the findings for this study. |

## **Data Protection**

The personal information we collect and use to conduct this research will be processed in accordance with UK data protection law as explained in the Participant Information Sheet and the <a href="Privacy Notice for Research Participants">Privacy Notice for Research Participants</a>.

By signing this consent form, I declare that I have provided accurate identity details (full name and electronic signature).

| Name of Participant | Signature | <br>Date |
|-----------------------------------|-----------|----------|
| Name of Participant | Signature | Date |
| Name of the person taking consent | Signature | Date |

Both the participant and the research team will keep an electronic copy of the above completed consent form.